CLINICAL TRIAL: NCT05982041
Title: A Prospective Cohort Study to Identify a Stratified Approach in the Diagnosis, Treatment in Adult Idiopathic Inflammatory Myopathy With Cardiac Injury
Brief Title: Adult Idiopathic Inflammatory Myopathy With Cardiac Injury
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Wang Qiang, The First Affiliated Hospital with Nanjing Medical University, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: IIMCI-1
Record Dates: First submitted 2023-07-01; First posted 2023-08-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Myopathy; Cardiac Disease
MeSH Terms: conditions — Myositis; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- idiopathic inflammatory myopathy

SUMMARY:
Adult patients with suspected or confirmed idiopathic inflammatory myopathy (IIM) will be recruited. Patients will be approached, consented, have baseline demographics, diagnostics and disease activity measures recorded, and blood taken. The collection of data and biological material will mirror usual clinical practice as far as possible. Subjects will ideally attend further visits at 3, 6 and 12 months to have bloods taken, outcome measures recorded and questionnaires completed.In addition, blood, muscle biopsies and imaging undertaken as part of usual care will also be collected for research purposes to measure a number of biomarkers for the assessment of diagnostic accuracy and clinical utility evaluation. As per usual practice, a muscle biopsy will be performed at baseline, and a further biopsy offered at 6 months to assess treatment response. A magnetic resonance (MR) muscle protocol will also be performed as per usual clinical practice, and a gadolinium-enhanced MR heart scan offered. Both these scans will be repeated at 6-12 months. An existing electronic database entry system will be used for data entry and capture on an anonymised basis.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had a confirmed (muscular biopsy, electromyogram, magnetic resonance imaging) or suspected clinically myositis
* Age over 18 years old
* Signature of the informed consent form for the study

Exclusion Criteria:

* Patients with disease duration >2 years
* Patients < 18 years
* Confirmed non-inflammatory myopathies
* Myositis secondary to alcohol or drug abuse
* Patients unwilling or unable to give consent
* Patients with poor or no venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a confirmed or suspected myositis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2033-01-01 (Estimated); Study Completion 2043-01-01 (Estimated)

PRIMARY OUTCOMES:
The emergence of late gadolinium enhancement (LGE) positive in the different myositis subgroups based on radiological evaluations | 20 years
  On the basis of the late gadolinium enhancement (LGE) positive by CMR
The emergence of extra-cellular volume (ECV) > 30% in the different myositis subgroups based on radiological evaluations | 20 years
  On the basis of extra-cellular volume (ECV) > 30% by CMR

SECONDARY OUTCOMES:
Number of participants with a significant change levels of diagnostic biomarkers | 20 years
  This will depend on the specific biomarker/cytokine being measured
Differences in frequency of genetic variants associated with IIM and subtypes compared to population matched controls | 20 years
  Specific identified genetic variants will be identified as part of large scale genetic studies
Incidence of major cardio-vascular events | 20 years

IPD SHARING:
Plan to Share IPD: No